CLINICAL TRIAL: NCT06697990
Title: Exploring the Mechanism of Cerebrospinal Fluid Immune Microenvironment in Patients With Advanced Anaplastic Lymphoma Kinase (ALK)-Positive Lung Cancer With Brain Metastases Treated With Iruplinalib: an Interventional Study
Brief Title: Cerebrospinal Fluid Immune Microenvironment Mechanism in Anaplastic Lymphoma Kinase Positive Lung Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-NSCLC-IIT-001
Record Dates: First submitted 2024-10-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iruplinalib (Experimental): The treatment will be administrated for 16 weeks, after which the treatment regimen was determined by the investigator.
  Interventions: Drug: Iruplinalib

INTERVENTIONS:
Drug: Iruplinalib — 60 mg of Iruplinalib, once daily for 7 days, followed by 180 mg of Iruplinalib, once daily in a 28-days cycle.
  Other Names: WX-0593

SUMMARY:
This is an an interventional study to explore the mechanism of cerebrospinal fluid immune microenvironment in patients with advanced anaplastic lymphoma kinase (ALK)-positive non-small cell lung cancer with brain metastases treated with Iruplinalib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced non-small cell lung cancer(NSCLC) that is anaplastic lymphoma kinase (ALK)-postive as assessed by the next-generation sequencing (NGS) test.
* Confirmed diagnosis of brain metastases or suspected brain metastases
* Iruplinalib is proposed for treatment
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0-1
* Adequate organ and marrow function

Exclusion Criteria:

* Have serious gastrointestinal disease or other uncontrolled internal diseases and infections
* The presence of mental illness or substance abuse at the time of screening that may have affected compliance with the trial
* The presence of pleural fluid or ascites that requires treatment or is judged by the investigator to be uncontrollable at the time of screening
* Arterial/venous thrombosis events occurred within 6 months prior to administration, such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid levels of Immune cells,inflammatory cytokines,immunoglobulins and cell adhesion molecules | 28 days
  Cerebrospinal fluid levels of natural killer (NK) cells,CD3+ T cells,CD4+ T cells,CD8+ T cells,tumour necrosis factor alpha(TNF-α), interleukin-6(IL-6), interferon-gamma(IFN-γ), high C-reactive protein(hs-CRP),immunoglobulin A(IgA),immunoglobulin E(IgE),immunoglobulin G(IgG),immunoglobulin M(IgM),intercellular adhesion molecule 1(ICAM-1) and vascular cell adhesion molecule 1(VCAM-1).

SECONDARY OUTCOMES:
Iruplinalib concentration in cerebrospinal fluid | Day 28
  Iruplinalib concentration in cerebrospinal fluid.
Objective response rate | 16 weeks
  Objective response rate is defined as the percentage of participants who have a complete response or partial response.
Disease control rate | 16 weeks
  Disease control rate is defined as the percentage of participants who have a best overall response of complete response, partial response, or stable disease.
Intracranial objective response rate | 16 weeks
  Intracranial objective response rate is defined as above for objective Response Rate but it is only based on intracranial disease in the subset of patients with intracranial lesion.
Intracranial disease control rate | 16 weeks
  Intracranial disease control rate is defined as above for disease control rate but it is only based on intracranial disease in the subset of patients with intracranial lesion.